CLINICAL TRIAL: NCT01597427
Title: Intravenous Clonidine Does Not Reduce Pulmonary Artery Pressure in Patients Subjected to Cardiac
Brief Title: Reduction of Pulmonary Artery Pressure in Patients Subjected to Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Fernando dos Reis Falcao, Clinical Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNIFESP-02
Record Dates: First submitted 2012-05-08; First posted 2012-05-14 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Anesthesia
Keywords: Clonidine; Hypertension Pulmonary; Cardiac Surgical Procedures
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine (Sham Comparator): Administration of 2 μg/kg of intravenous clonidine.
  Interventions: Drug: Clonidine
- Placebo (Placebo Comparator): Injection of placebo solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — Administration of 2 μg/kg of intravenous clonidine
  Arms: Clonidine
Drug: Placebo — Injection of placebo solution.
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the ability of clonidine to reduce the mean pulmonary artery pressure in patients with pulmonary hypertension subjected to cardiac surgery.

DETAILED DESCRIPTION:
Prospective, clinical-interventionist, randomized, and double-blind study. Patients with group 2 pulmonary hypertension will be included and subjected to cardiac surgery with extracorporeal circulation. Mean pulmonary artery pressure and the doses of dobutamine and sodium nitroprusside will be assessed four times: before (T0) administration of 2 μg/kg of intravenous clonidine or a placebo, 30 minutes after the onset of treatment (T1), immediately after extracorporeal circulation (T2), and 10 minutes after the injection of protamine (T3).

ELIGIBILITY:
Inclusion Criteria:

* Signing an informed consent form,
* Aged 18 to 80 years
* Pulmonary hypertension due to left heart disease,
* Physical status 2 or 3 according to the classification system of the American Society of Anesthesiologists,
* Subjected to cardiac circulation with extracorporeal circulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduction pulmonary artery pressure | During intraoperative (hours)
  Assessed four times: before (T0) administration of 2 μg·kg-1 of intravenous clonidine or a placebo, 30 minutes after the onset of treatment (T1), immediately after ECC (T2), and 10 minutes after the injection of protamine (T3).

SECONDARY OUTCOMES:
Doses of Dobutamine | During intraoperative (hours)
  Evaluate the need for using and dose of dobutamine immediately after extracorporeal circulation between groups.
Doses of Sodium nitroprusside | During intraoperative (hours)
  Evaluate the need for using and dose of sodium nitroprusside immediately after extracorporeal circulation between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Fernando R Falcao, Ph.D., Study Chair — Federal University of São Paulo; Benedito B Joao, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Luiz Fernando dos Reis Falcao, São Paulo, São Paulo, Brazil